CLINICAL TRIAL: NCT06755762
Title: Using A Three-dimentional Culture Model for Circulating Tumor Cells Combined With Molecular Bioassays in Patients With Head and Neck Cancer to Help Determine the Precise Choice of Systemic Drugs to Improve Survival Outcomes
Brief Title: Using a 3D Culture Model for Circulating Tumor Cells Combined With Molecular Bioassays in Patients With HNSCC Cancer
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jason Chia-Hsun Hsieh, Professor Attending Physicians, Chang Gung Memorial Hospital
Other Study IDs: 202301979B0
Record Dates: First submitted 2024-12-04; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Circulating Tumor Cell; HNSCC
Keywords: circulating tumor cell; organoid; HNSCC
MeSH Terms: conditions — Neoplastic Cells, Circulating; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Genomic DNA was isolated from blood to control for germline variants using the DNeasy Blood and Tissue Kit.Biallelic drop out was calculated from germline heterozygous single-nucleotide polymorphisms (SNPs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: healthy donors
  Interventions: Other: Organoid 3D culture
- experimental: HNSCC patients
  Interventions: Other: Organoid 3D culture

INTERVENTIONS:
Other: Organoid 3D culture — Investigate different normal cells (lung, bone, soft tissue, liver, etc) as metastatic organs to simulate the behaviors of CTCs in metastatic sites
  Other Names: without cancer patients

SUMMARY:
Cancer has been a significant cause of human death in the recent two decades, although detection, diagnosis, and cancer treatments improved and evolved rapidly. Till now, the reasons why some cancer recurs and others do not remain unclear. Since 2004, circulating tumor cell (CTC) has been well-recognized that CTCs in the circulatory system are associated with cancer metastasis. The fundamental studies of CTCs hold tremendous potentials for probing the biological insights on the molecular mechanisms underlying cancer metastasis, cancer-related gene mutation, or biomarker discovery. However, the low purity (one of the natural limitations) of isolated samples often hampered CTC-directed studies' utility. For that, investigators used a well-established device (ODEP, optically-induced-dielectrophoresis) to isolate viable and high-purity CTCs for the following investigations. Investigators team developed a protocol in the past months and succeeded in cultivating CTCs (near 100%) for further drug tests and had a technology platform of organoid culture system developing in 2020. The preliminary results of the experiments showed a promising combination. That urges investigators to propose a 3-year project investigating CTC culture in the organoid system to look at (1) the behavior of CTCs in organ cell background (organoid), (2) the influences of different background cells, (3) the different in-vitro (or in-organoid) response of CTCs to specific drugs (pembrolizumab, nivolumab, cetuximab, cisplatin, 5-FU, taxanes) of head and neck squamous cell carcinoma. In the meantime, investigators will look at the genomic alterations of those CTCs growing fast and well in the organoid systems to find possible precipitating metastasis genes at a scale of cell (CTC) level. Investigators believe that the project is doable and possibly help human cancer control and understanding.

DETAILED DESCRIPTION:
Strikingly, accounting for 7.6 million deaths (around 13% of all deaths) in 2008, cancer is a leading cause of death worldwide, according to the statistical data from the World Health Organization (WHO). WHO also estimates 12 million cancer deaths worldwide in 2030. More than 285,000 people every year are diagnosed with cancer in the United Kingdom, and the current estimate is that more than one in three people will develop a form of cancer at some point in their lifetime . In Taiwan, cancer is also one of the major causes of death in the Taiwanese population according to the statistical data from the Department of Health (Taiwan). The expense associated with cancer patient care and therapy is high, and is a burden for the family of cancer patients. Hence, cancer not only is a huge threat for human life, but also has a serious social impact and national health. Fighting cancer is therefore one of the priority tasks in biomedical research. Cancer is a generic term for a large group of diseases that can affect any part of the body. Other terms used are malignant tumors and neoplasms. One defining feature of cancer is the rapid creation of abnormal cells that grow beyond their usual boundaries, and which can then invade adjoining parts of the body and spread to other organs . This process is referred to as metastasis. A primary cancer is a tumor mass present at the site of initial conversion of a normal cell to a tumor cell. If all cells remained in the primary tumor, cancer would be of little clinical importance. Growth of the tumor would produce pressure on surrounding tissue, but the well-defined tumor mass could be excised by surgery in a straightforward and permanent way. Nevertheless, tumor cells do not always remain at the primary site but move away by one of two processes: (a) invasion, or the movement of cells into neighboring space occupied by other tissues; and (b) metastasis, the spread of cells to areas not directly adjacent to the primary tumor usually via the bloodstream, lymphatic system, or through body space. Metastasis generally occurs in several stages: (c) detachment of cells from the primary tumor, (2) penetration and migration of tumor cells into lymph vessels or blood vessels, (3) lodging of tumor cells in blood vessels of distant organs, (d) invasion of tumor cells through the vessels walls and into the tissue of secondary sites, (e) growth of secondary tumors at the secondary sites . Cancer metastasis is a leading cause of cancer-derived lethality .

Circulating tumor cells (CTCs) are the rare cell species present in the peripheral blood that has been documented since 1869. It is well recognized that the presence of CTCs in the circulatory system is associated with cancer metastasis. The fundamental studies of CTCs hold tremendous potentials for probing the biological insights on the molecular mechanisms underlying cancer metastasis, cancer-related gene mutation[8], or biomarker discovery, which could both facilitate and accelerate scientists to develop new therapeutic solutions for future cancer care. In addition, the CTCs in blood circulation are thought to be mainly responsible for cancer progression or relapse , and thus are obvious targets of cancer therapy. Several emerging studies have showed that CTCs can be a real-time tumor biopsy that can be utilized in new drug development , and the selection of therapeutic regimens, by which the pharmacodynamics or clinical response of CTCs to the treatments can be established, respectively. For the latter clinical utility, the responses of CTCs to chemotherapy (e.g. drug sensitivity or resistance) not only can be used to guide the personalized cancer chemotherapy but also can be a clinically important indicator for monitoring long-term therapeutic efficacy, disease recurrence, and the change of biological characteristics of CTCs in a real time and noninvasive manner. This can provide predictive information for the adjustment of therapeutic scheme throughout the stages of cancer care. However, to the best of investigators knowledge, the use of CTCs has been limited mainly because of its rarity with an approximate concentration of 1 CTC per 105 -107 blood mononuclear cells, and such rarity nature makes it difficult both to detect and isolate. Moreover, investigators understanding of their biological or chemico-physical properties has been limited by the availability of technologies capable of isolating them in sufficient numbers. The amount of isolated CTCs is too low to reach the lowest sample limits of many detailed molecular and functional experiments. These factors resulting from low recovery rates slow down the clinical use of CTCs. Despite the limitations of current CTC-isolating methods, circulating cancer cells have been detected in a vast majority of epithelial cancers, such as breast, prostate, lung, and colon cancers. Patients with metastatic lesions are tended to have CTCs detected in their blood; however, these have also been reported in some localized cancers. Therefore, for further detailed researches, characteristics of CTCs and mechanism of distant metastasis, developing a reliable, high recovery rate with high purity of isolated CTCs is currently most challenging and critical.

Precision medicine is a relatively new strategy to identify the best therapy for each patient's disease, based on the genomic characterization of an individual's tumor, and while this approach holds tremendous promise, the complex genetic and epigenetic profiles of individual tumor cells has made this approach challenging. Another approach to predicting treatment response has been to directly test tumor cells from patients in established two-dimensional (2D) models in drug screening studies. Recent studies by Yoshii and colleagues indicated that three-dimensional (3D) culture conditions may be more reflective of tumor in vivo growth conditions than 2D cell cultures. To explore this, we have previously established a 3D culture models for HNSCC and compared to 2D cultures and in vivo tumors models.

Patient-derived xenografts (PDXs) have been widely used for drug screening studies to overcome the limitations of 2D screening studies. However, PDX models also have some limitations; including, low engraftment rates of cancer in nude mice, striking differences in pharmacokinetics between two humans and mice, and the lengthy time required for drug screening (4-8 months) studies in PDXs. Recently, 3D cell culture models have been used for drug screening studies and biomarker analysis. Establishment of cell lines from 2D cultures of tumors derived from patient tissue has a low success rate, and only select tumor cells can survive in the 2D environment which may be reflected in an altered tumor heterogeneity from the original tumor. Furthermore, it is well known that long term culture can select for genetic alterations. Since most 3D culture models derived from established 2D cell lines do not maintain the original tumor phenotype, development of 3D cancer organoid cultures directly from a patient's cancer tissue which includes cancer stem cells, can better recapitulate the character of the patient's tumor than those derived from cells previously passaged as 2D cultures. Although, there are published methods to generate cancer organoid in various cancer types, establishment of HNSCC cancer organoids has not been attempted. Therefore, investigators were interested to develop a HNSCC cancer organoid model and characterizes it properties and compare them to features of the original.

The Cancer Tissue-Originated Spheroids (CTOS) method is a technique to establish cancer organoid lines reported by Kondo et al. which showed highly established rate in colon cancer, lung cancer and bladder cancer. In this method, the cell lines obtained are cultured and maintained as organoids. Organoids have the capabilities to maintain the same histological features of the original tumors. In addition, the population of cancer stem cell is very similar between the original tumor and organoids lines, indicating that the CTOS method can recapitulate the character of the original tumor. In this proposal, investigators attempt to evaluate the feasibility of establishment and characterization of HNSCC organoids, and the utility of these cell lines as a model for drug screening and testing.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18
2. agree with blood drawing and follow the procedure of the trial

a.health participants:without cancer over 5 yaers b.cancer participants:pathology: metastatic HNSCC patients

Exclusion Criteria:

1. health participants:with serious illness
2. cancer participants:none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Develop the CTC culture system (isolated by negative selection strategy and ODEP platform) and organoid 3D culture system for CTC from health participants and HNSCC cancer participants.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
cell density and numbers | baseline
  CTC number low(<10) and high(>100)
cytokines detection-EpCAM | baseline
  For negative selection of CTCs by the negative selection system.To deplete EpCAM leukocytes, a EpCAM depletion cocktail was mixed with the collected nucleated cells
cytokines detection-CD-45+ leukocytes | baseline
  For negative selection of CTCs by the negative selection system.To deplete CD-45+ leukocytes, a CD-45 depletion cocktail was mixed with the collected nucleated cells
counting of EpiCAM-positive and Hoechst-positive cells | baseline
  Positive Selection method.The cell recovery is determined by counting EpiCAM-positive and Hoechst-positive cells under microscope with hemocytometer. Human samples will go through the whole processes without spiking steps

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, PhD, Study Chair — Division of Oncology, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan